CLINICAL TRIAL: NCT06739993
Title: Effects of Autonomic Nervous System Modulation by Heart Rate Variability Biofeedback Training With Resonant Frequency Breathing on Glucose Metabolism in Individuals With Prediabetes
Acronym: RwHRVBFinPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Benedict Herhaus, Ph.D., Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-16489; 540546352 (Other Grant/Funding Number: Deutsche Forschungsgemeinschaft (DFG, German Research Foundation))
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Prediabetes
Keywords: prediabetes; glucose metabolism; heart rate variability-biofeedback training; resonance frequency breathing; oral glucose tolerance test
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Intervention Model Description: Randomized-controlled Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Resonance frequency breathing with heart rate variability biofeedback training (RFB-HRV-BF) (Experimental): The mobile system "eSense Pulse" by Mindfield Biosystems Ltd. (Gronau, Germany) was used for RFB-HRV-BF training. The participants sat in an upright position, started the training via the eSense app on their smartphone, and were instructed to practice breathing at their individually determined resonance frequency.During training, a ball that expands (breathe in) and shrinks (breathe out) on the screen specified the breathing frequency goal to a value of six cycles per minute (five seconds inspiration, five seconds expiration). The HRV was visualized by new symbols varying in color depending on the respectively measured values, which appeared every ten seconds.
  Interventions: Behavioral: Resonance frequency breathing with heart rate variability biofeedback training
- Anti-Stress program (Active Comparator): The mobile system eSense Pulse from Mindfield Biosystems is used for the digital anti-stress program. To do this, the participants put on a chest strap with a sensor and can start training via the eSense app. The anti-stress program is carried out using a procedure generated for the study. During the anti-stress program units, the participants receive application-related information and tips to better understand the topic of stress, identify stressors in their own lives and reduce stress. The active control intervention of the anti-stress program was selected to investigate the effect of a specific stress level reduction without the direct modulation of physiological mechanisms of action as with HRV-BF-RFA.
  Interventions: Behavioral: Anti-Stress program

INTERVENTIONS:
Behavioral: Resonance frequency breathing with heart rate variability biofeedback training — During training, a ball that expands (breathe in) and shrinks (breathe out) on the screen specified the breathing frequency goal to a value of six cycles per minute (five seconds inspiration, five seconds expiration). The HRV was visualized by new symbols varying in color depending on the respectively measured values, which appeared every ten seconds. When the participants achieved the specified breathing frequency, resulting in an increased sinus arrhythmia, the symbols appearing on the smartphone display were green. When the participants did not achieve the specified breathing frequency, the symbols appeared in yellow (non-significant deviation), orange (significant deviation), or red (very significant deviation). The participants were instructed to adjust their breathing frequency to reach emergence of as many green symbols as possible for the entire training session.
  Other Names: RFB-HRV-BF
  Arms: Resonance frequency breathing with heart rate variability biofeedback training (RFB-HRV-BF)
Behavioral: Anti-Stress program — The mobile system eSense Pulse from Mindfield Biosystems is used for the digital anti-stress program. To do this, the participants put on a chest strap with a sensor and can start training via the eSense app. The anti-stress program is carried out using a procedure generated for the study. During the anti-stress program units, the participants receive application-related information and tips to better understand the topic of stress, identify stressors in their own lives and reduce stress. The active control intervention of the anti-stress program was selected to investigate the effect of a specific stress level reduction without the direct modulation of physiological mechanisms of action as with HRV-BF-RFA.
  Other Names: ASP
  Arms: Anti-Stress program

SUMMARY:
Approximately 20% of adults have prediabetes in Germany. Prediabetes is defined as a condition with glucose levels outside the normal range but not yet meeting the criteria for type 2 diabetes. The pathogenesis of prediabetes, as well as of type 2 diabetes, involves whole-body insulin resistance associated with inadequate insulin secretion. These two central processes of glucose regulation are modulated by the brain. The brain communicates via the autonomic nervous system (ANS) with metabolically important organs in the periphery to modulate insulin sensitivity and insulin secretion. These processes are impaired in individuals with prediabetes and diabetes. An ANS sympathovagal imbalance has also been observed in individuals with prediabetes. There are no specific therapeutic approaches to improve ANS sympathovagal imbalance. It is assumed that resonant frequency breathing (RFB) maximizes heart rate variability (HRV) through rhythmization of breathing, heartbeat, and blood pressure. Through this state of coherence, the activity of the parasympathetic nervous system is upregulated, and the activity of the sympathetic nervous system is suppressed, leading to an increase in modulation of ANS activity. Several studies have demonstrated that heart rate variability-biofeedback (HRV-BF) interventions improve HRV, reduce stress and anxiety, and alleviate symptoms in patients with various medical conditions. To the best of current knowledge, no study has investigated the effect of HRV-BF-RFB on glucose metabolism. Therefore, the proposed randomized controlled non-blinded trial aims to gain evidence about the effect of HRV-BF-RFB compared to an anti-stress program on glucose metabolism in individuals with prediabetes. Glucose metabolism is characterized using the 75 g oral glucose tolerance test. There are two potential mechanisms by which HRV-BF-RFB may improve glucose metabolism in individuals with prediabetes: (a) a 0°-phase relationship between heart oscillations and breathing, maximizing the amplitude of respiratory sinus arrhythmia (RSA), and (b) activation of the cholinergic anti-inflammatory pathway. The investigators hypothesized that in individuals with prediabetes, the HRV-BF-RFB intervention will improve glucose metabolism and glucose variability.

ELIGIBILITY:
Inclusion Criteria:

* Presence of prediabetes Fasting glucose: 100-125 mg/dl (5.6-6.9 mmol/L) and/or HbA1c in %: 5.7-6.4 (39-47 mmol/mol Hb) and/or 2-hour value of the 75 g OGTT: 140-199 mg/dl (7.8-11.0 mmol/L)

  * This is checked using a 75 g OGTT in a screening visit.
* Age between 18 and 65 years
* BMI between 20 and 40 kg/m²

Exclusion Criteria:

* Diabetes mellitus
* Malignant diseases within the last 5 years before randomization
* History of gastrointestinal surgery
* Pancreatic diseases other than pancreatic lipomatosis
* Acute diseases or infections
* Regular intake of cardiac drugs that affect heart rate within the last 4 weeks before the first measurement (e.g. beta-receptor blockers, antiarrhythmics, etc.)
* Intake of centrally acting drugs
* Medical contraindications to a meaningful interpretation of the heart rate analysis (e.g. patients with pacemakers, atrial fibrillation or other arrhythmias)
* Chronic diseases (particularly metabolic diseases, heart diseases, blood diseases)
* Endocrinological disease other than substituted hypothyroidism
* Mental illnesses
* Intake of drugs that can affect blood sugar metabolism (e.g. steroids)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Glucose metabolism | Baseline, four weeks, and eight weeks.
  Glucose metabolism was assessed through a frequently-sampled 75 g oral glucose tolerance test (OGTT) starting at 8:00 a.m. after an overnight fast. After basal blood sampling, the participants drank a 75 g glucose solution, with further blood samples taken at 30, 60, 90, and 120 minutes after glucose ingestion. Areas under the curve were calculated based on the trapezoid method.

SECONDARY OUTCOMES:
Glucose stimulated insulin secretion | Baseline, four weeks, and eight weeks.
  Glucose stimulated insulin secretion was assessed as oral Disposition Index and as ratio of the areas under the C-peptide curves and the areas under the glucose curves during the first 30 minutes of the OGTT (AUC C-peptid0-30/AUC glucose0-30). For the estimation of insulin sensitivity, HOMA-IR was used for the fasting state and Matsuda Index [29] for the post-glucose load situation. Insulin clearance was estimated by the ratio of the areas under the C-peptide and insulin curves during the OGTT (AUC C-peptide0-120/AUC insulin0-120).

OTHER OUTCOMES:
Interstitial fluid glucose levels in mg/dL | Two weeks before the intervention, two weeks after the intervention
  The daily profiles of the interstitial fluid glucose levels are recorded using continuous glucose measurement systems (FreeStyle Libre Pro iQ). These data enable the calculation of indices to assess glucose variability (standard deviation, coefficient of variation, MAGE index, MODD index) and glucose tolerance (daily mean values, AUC). Each measurement period lasted 14 days, as per the sensor lifespan.
Cytokines | Baseline, four weeks, and eight weeks.
  The cytokine profile is quantified using 48 analytes measured as a multiplex assay (proximity extension assay, Olink Proteomics, 2021). The 45 immune-related proteins (in pg/mL) are: IL-18, HGF, CCL19, CCL2, MMP12, LTA, FLT3LG, TNF, IL17A, IL2, ILF17F, CSF3, IL1B, OLR1, TNFSF12, CXCL10, VEGFA, IL33, TSLP, IFNG, CCL4, TGFA, IL13, CXCL8, CCL8, IL6, CCL13, CSF2, CCL7, IL4, TNFSF10, OSM, MMP1, EGF, IL7, IL15, CSF1, CXCL9, CXCL11, IL17C, CXCL12, CCL11, IL10, CCL3, EBI3_IL27.

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University Medical Center Mainz - Medical Psychology and Medical Sociology, Mainz, Mainz
  - University Medical Center of the Johannes-Gutenberg University, Department of Medical Psychology and Medical Sociology, Mainz, Rhineland-Palatinate

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Herhaus B, Thesing G, Conrad R, Petrowski K. Alterations in heart rate variability and pro-inflammatory cytokine TNF-alpha in individuals with panic disorder. Psychiatry Res. 2023 Apr;322:115107. doi: 10.1016/j.psychres.2023.115107. Epub 2023 Feb 12. PMID 36796202
- [Background] Herhaus B, Siepmann M, Kahaly GJ, Conrad R, Petrowski K. Effect of a Biofeedback Intervention on Heart Rate Variability in Individuals With Panic Disorder: A Randomized Controlled Trial. Psychosom Med. 2022 Feb-Mar 01;84(2):199-209. doi: 10.1097/PSY.0000000000001031. PMID 34654028
- [Background] Herhaus B, Kalin A, Gouveris H, Petrowski K. Mobile Heart Rate Variability Biofeedback Improves Autonomic Activation and Subjective Sleep Quality of Healthy Adults - A Pilot Study. Front Physiol. 2022 Feb 17;13:821741. doi: 10.3389/fphys.2022.821741. eCollection 2022. PMID 35250623
- [Background] Herhaus B, Conrad R, Petrowski K. Effect of a slow-paced breathing with heart rate variability biofeedback intervention on pro-inflammatory cytokines in individuals with panic disorder - A randomized controlled trial. J Affect Disord. 2023 Apr 1;326:132-138. doi: 10.1016/j.jad.2023.01.091. Epub 2023 Jan 28. PMID 36720404
- [Background] Heni M, Wagner R, Willmann C, Jaghutriz BA, Vosseler A, Kubler C, Hund V, Scheffler K, Peter A, Haring HU, Preissl H, Kullmann S, Fritsche A. Insulin Action in the Hypothalamus Increases Second-Phase Insulin Secretion in Humans. Neuroendocrinology. 2020;110(11-12):929-937. doi: 10.1159/000504551. Epub 2019 Nov 5. PMID 31689708
- [Background] Heni M, Wagner R, Kullmann S, Veit R, Mat Husin H, Linder K, Benkendorff C, Peter A, Stefan N, Haring HU, Preissl H, Fritsche A. Central insulin administration improves whole-body insulin sensitivity via hypothalamus and parasympathetic outputs in men. Diabetes. 2014 Dec;63(12):4083-8. doi: 10.2337/db14-0477. Epub 2014 Jul 15. PMID 25028522
- [Background] Heni M, Wagner R, Kullmann S, Gancheva S, Roden M, Peter A, Stefan N, Preissl H, Haring HU, Fritsche A. Hypothalamic and Striatal Insulin Action Suppresses Endogenous Glucose Production and May Stimulate Glucose Uptake During Hyperinsulinemia in Lean but Not in Overweight Men. Diabetes. 2017 Jul;66(7):1797-1806. doi: 10.2337/db16-1380. Epub 2017 Feb 7. PMID 28174292